CLINICAL TRIAL: NCT00809237
Title: A Phase II With a Lead in Phase I Study to Examine the Tolerability, Safety Profile and Efficacy of Hydroxychloroquine and Gefitinib in Advanced Non-Small Cell Lung Cancer
Brief Title: Hydroxychloroquine and Gefitinib to Treat Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Massachusetts General Hospital (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Chin Tan Min, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS 01/03/08; 2008/00196 (Other: NHG Doman Specific Review Board)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Gefitinib; Hydroxychloroquine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib, Hydroxychloroquine (Experimental): For the lead in phase I study, recruited patients will receive one week of 250 mg of Gefitinib, before HCQ at the assigned dose is introduced in addition to Gefitinib 250 mg om.
  After the MTD of HCQ is determined, the phase II study will proceed with the combination of 250 mg of Gefitinib and the MTD dose of HCQ.
  Interventions: Drug: Gefitinib, Hydroxychloroquine

INTERVENTIONS:
Drug: Gefitinib, Hydroxychloroquine — Gefitinib 250 mg om Hydroxychloroquine at maximally tolerated dose
  Other Names: Iressa

SUMMARY:
Non-small cell lung cancer (NSCLC) is the most common cause of cancer mortality in men and women in Singapore.Chemotherapy and biologically targeted agents can extend survival only modestly for these patients; therefore, discovery of novel ways to prolong the disease course is a top research priority.

The epidermal growth factor receptor (EGFR) signaling pathway plays a central role in the neoplastic transformation of NSCLC and promotes cancer cell survival, metastasis, and angiogenesis. The predominance of EGFR signaling in NSCLC makes the pathway an attractive candidate for the development of targeted therapeutics. Over the last three years, the FDA has approved two drugs for salvage treatment of NSCLC, gefitinib (Iressa ®, formerly known as ZD1839) and erlotinib (Tarceva ®, formerly known as OSI-774). Both are small molecule orally-bioavailable tyrosine kinase inhibitors (TKIs) of the EGFR TK domain, and have been shown to improve survival compared to placebo in asian patients when administered after failure of first or second line chemotherapy for advanced NSCLC.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the most common cause of cancer mortality in men and women in Singapore.Chemotherapy and biologically targeted agents can extend survival only modestly for these patients; therefore, discovery of novel ways to prolong the disease course is a top research priority.

The epidermal growth factor receptor (EGFR) signaling pathway plays a central role in the neoplastic transformation of NSCLC and promotes cancer cell survival, metastasis, and angiogenesis. The predominance of EGFR signaling in NSCLC makes the pathway an attractive candidate for the development of targeted therapeutics. Over the last three years, the FDA has approved two drugs for salvage treatment of NSCLC, gefitinib (Iressa ®, formerly known as ZD1839) and erlotinib (Tarceva ®, formerly known as OSI-774). Both are small molecule orally-bioavailable tyrosine kinase inhibitors (TKIs) of the EGFR TK domain, and have been shown to improve survival compared to placebo in asian patients when administered after failure of first or second line chemotherapy for advanced NSCLC.

Recently, it was found that somatic mutations in the EGFR gene sensitize NSCLC tumors to TKIs. These mutations are present in approximately 50 % of asian patients with NSCLC. Retrospective studies suggest that patients harboring a mutation may derive greater clinical benefit from treatment with TKIs than patients without a mutation.

Nevertheless, all patients that benefit from TKI treatment ultimately develop resistance to therapy manifesting as progression of their cancer, after which there remains few, if any treatment options. Hence, there would be vast clinical utility in understanding the mechanisms of TKI resistance and developing strategies to reverse or prevent it.

We have preliminary data which shows that the combination of hydroxychloroquine and gefitinib results in delayed acquired resistance to gefitinib in cell lines that harbour the EGFR mutation. In addition, the addition of hydroxychloroquine to gefitinib can result in reversal of acquired resistance to gefitinib. Much parallel has been observed in resistance mechanisms between NSCLC cell lines and molecular changes observed in patients thus far.

The long term aim therefore is to examine the efficacy of this combination in delaying acquired resistance to gefitinib in NSCLC patients.

First, however, the MTD and DLT of each drug when used in combination therapy will be examined in this study. The other aim is to examine the pharmacokinetic effect and interactions of hydroxychloroquine on gefitinib, and vice versa. Gefitinib is usually well tolerated, with main toxicities of rash and diarrhoea. Hydroxychloroquine is also FDA approved and widely used and generally well-tolerated for rheumatological conditions.

ELIGIBILITY:
Inclusion Criteria:

For the lead in phase I study:

1. Pathologically confirmed diagnosis of non-small cell lung cancer.
2. Stage IIIB with pleural effusion or stage IV disease by the American Joint Committee on Cancer (AJCC) 6th edition staging criteria.
3. Age equal to or greater than 21 years
4. Measurable disease, defined according to RECIST criteria
5. Performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group(ECOG) Performance Status scale.
6. At least 2 weeks since prior radiation treatment, chemotherapy or targeted therapy (from the day that protocol treatment begins).

   Patients who had been on gefitinib should have a wash out period of two weeks prior to commencement of treatment drugs for this study.
7. Adequate organ function including the following:

   * Adequate bone marrow reserve:

     * Total white blood cell count (WBC) > 3.0 x 109/L
     * Platelet count >100 x 109/L
     * Hemoglobin >8 g/dL
   * Hepatic:

     * Bilirubin: = 1.25 times the upper limit of normal (ULN)
     * Alanine transaminase (ALT): = <5 times the ULN
     * Aspartate transaminase (AST): = <5 times the ULN
   * Renal: Serum creatinine =< 1.5 times the ULN, or creatinine clearance =>60mL/minute as calculated by the standard Cockcroft Gault formula.
8. Approval for HCQ treatment by an eye doctor, based on a screening eye exam. Examples of disqualifying baseline conditions include macular degeneration and other retinal disease, see exclusion criteria.
9. Willingness to comply with protocol procedures including the blood-sampling schedule for PK analyses and periodic eye examinations.
10. Willingness to participate in clinical research as evidenced by their signature on the informed consent form.
11. Tumor block from subject's biopsy or surgical resection specimen should ideally be available but is not a mandatory requirement for study entry.

For the phase II study:

Inclusion criteria as above, except that:

1. NSCLC patients must be non-smokers and have adenocarcinomas.
2. Patients who had been on gefitinib should have a wash out period of two weeks prior to commencement of treatment drugs for this study. They must have responded to Gefitinib previously (either CR, PR or SD) for more than twelve weeks to be eligible.

Exclusion Criteria:

For both lead in phase I and phase II study:

1. Current use of hydroxychloroquine for any reason.
2. Known hypersensitivity to chloroquine, hydroxychloroquine, or any closely related drug.
3. Known hypersensitivity to erlotinib, gefitinib, or any closely related drug.
4. Glucose-6-phosphate dehydrogenase (G6PD) deficiency, as HCQ may cause hemolytic anemia in patients with G6PD deficiency.
5. Cataracts that would interfere with required funduscopic examinations, or severe baseline visual impairment including macular degeneration, retinopathy or visual field changes, or having only one functional eye. All patients must undergo a screening eye exam prior to enrollment.
6. Pregnant or breastfeeding. HCQ crosses the placenta and use is not recommended during pregnancy except for life-threatening malaria. The effects of gefitinib on a fetus are unknown. For these reasons, female subjects of childbearing age must practice acceptable methods of birth control to avoid pregnancy. Male subjects must also practice acceptable methods of birth control to prevent pregnancy of a partner.
7. Symptomatic CNS metastases or newly diagnosed CNS metastases that have not yet been definitively treated with radiation and/or surgery. Note that patients with a history of CNS metastases or cord compression are allowable if they have been definitively treated and are clinically stable. Maintenance steroids are allowed but maintenance seizure medication is not allowed.
8. Prior radiation therapy inclusive of all identified target lesions. Note that prior palliative radiation to bony disease, CNS disease, or a limited thoracic area is allowed, provided that there is measurable disease outside the field and radiation is completed at least two weeks prior to starting treatment and the patient has fully recovered from all side effects.
9. Any evidence of clinically active interstitial lung disease. Note that patients with chronic, stable radiographic changes who are asymptomatic need not be excluded.
10. Malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
11. Although not an absolute exclusion criteria, caution should be exercised in patients with a diagnosis of prophyria or non-light-sensitive psoriasis, as HCQ can significantly exacerbate both of these conditions.
12. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study, in the opinion of the investigator.
13. Use of any non-FDA approved or investigational agent within 2 weeks of enrolling onto the trial, or failure to recover from the side effects of any of these agents.
14. Penicillamine use for Wilson's disease or any other indication, as concomitant use with HCQ can increase toxicity to penicillamine.
15. Concommitant use of anti-convulsants is not allowed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
For the phase I lead in study: To identify the tolerability, the dose limiting toxicity (DLT) and the general safety profile of HCQ and gefitinib when used in combination. | 2 years
For the phase II study: To determine the response rates to HCQ and Gefitinib. | 2 years

SECONDARY OUTCOMES:
For the phase I lead in study: To determine the PK (pharmacokinetic) parameters of HCQ plus gefitinib. | 2 years
For the phase II study: To determine the time to progression for patients treated with HCQ and Gefitinib. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tan Min Chin, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore